CLINICAL TRIAL: NCT04389437
Title: OCT-Angiography and Adaptive Optics in Patients With Memory Impairment
Acronym: OCTAVO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AMR_2020_3
Record Dates: First submitted 2020-05-12; First posted 2020-05-15 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Amnesia; Alzheimer Disease; Lewy Body Disease; Parkinsons Disease With Dementia
Keywords: OCT-A; adaptative optics
MeSH Terms: conditions — Amnesia; Alzheimer Disease; Lewy Body Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- NCD patients (case) (Experimental): Patient diagnosed with Alzheimer's disease or parkinsonian dementia / Lewy body dementia or other mild or severe NCD defined by international criteria.
  Interventions: Procedure: Ophthalmological exam; Procedure: Blood pressure measurement
- Control patients with memory complaint (Other): Normal neuropsychological evaluation during assessment
  Interventions: Procedure: Ophthalmological exam; Procedure: Blood pressure measurement
- Control patients without memory complaint (Other): MMS score and / or the Montreal Cognitive Assessment grid (MoCA) ≥26 / 30, No memory complaint
  Interventions: Procedure: Ophthalmological exam; Procedure: Blood pressure measurement

INTERVENTIONS:
Procedure: Ophthalmological exam — OCT-A and AO
Procedure: Blood pressure measurement — Blood pressure measurement before the ophthalmological exam

SUMMARY:
Studies suggest an association between retinal abnormalities and NCD (Neuro Cognitive Disorders) whether they are linked to proven or prodromal Alzheimer's disease (aMCI : amnestic mild cognitive impairment), or to other neurodegenerative diseases such as frontotemporal dementia or Lewy body diseases.

These retinal anomalies objectified by OCT-A (Optical coherence tomography angiography) and adaptive optics (AO) appear different depending on the pathologies and could therefore serve as markers in vivo of the pathophysiological processes underlying NCD.

No study to date has studied the retina and its vessels in NCD using adaptive optics. In this pilot study, we are proposing a combination of two new ophthalmological imaging techniques (OCT-A and AO), which allow rapid in vivo analysis in a completely non-invasive way of the morphology of small vessels as well as architecture of the retina to better specify the retinal anomalies associated with NCD. We will compare the parameters in OCT-A and AO between patients with NCD and controls without NCD (with memory complaint or without) and will seek to determine if there are different profiles according to the causes of NCD.

ELIGIBILITY:
Inclusion Criteria:

* Patient presenting in memory consultation for memory complaint or person accompanying a patient in memory consultation for memory complaint

Exclusion Criteria:

* pregnant or lactating women
* history of known non-degenerative neurological pathology (tumor, stroke territorial, in particular multiple sclerosis)
* history of retinal pathology
* ametropia greater in absolute value than 3 diopters on the sphere, or/and 1.5 diopters on the cylinder.
* history of taking ethambutol for more than 2 months
* history of takingsynthetic antimalarial for more than 2 years
* Mini Mental State Score (MMS) and / or Montreal Cognitive Assessment (MoCA) <10 for patients and 26 for accompanying persons
* MRI contraindication (for patients only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2020-06-26 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Wall to lumen ratio (WLR) | Baseline (Inclusion)
  Measured in adaptive optics, compared between patients case with NCD and patient controls without NDC found

CONTACTS AND LOCATIONS:
Overall Officials: Antoine MOULIGNIER, MD, Principal Investigator — Fondation A. de Rothschild
Locations (1):
- Hôpital Fondation A. de Rothschild, Paris, France